CLINICAL TRIAL: NCT01162785
Title: Phase 1B Intravesical Administration of SCH 721015 (Ad-IFNa) in Admixture With SCH 209702 (Syn3) for The Treatment of BCG Refractory Superficial Bladder Cancer
Brief Title: 1B Intravesical Administration of SCH 721015 (Ad-IFNa) in Admixture With SCH 209702 (Syn3) for The Treatment of BCG Refractory Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: FKD Therapies Oy of Finland (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0938; P50CA091846 (NIH); NCI-2010-01769 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Bladder Cancer
Keywords: BCG Refractory Superficial Bladder Cancer; SCH 721015; Syn3; novel excipient; interferon -alpha-2b; Intravesical; urine IFNa; transitional cell carcinoma of the bladder; superficial non-muscle invasive tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Dose SCH 721015 (Experimental): Part1: 2 Instillations of intravesical SCH 721015 (on Day 1 and 4) at a dose concentration of 3x1011particles/mL given in a 75 mL total volume
  Interventions: Drug: SCH 721015
- Second Dose SCH 721015 (Experimental): Part 2: Subjects who have a complete response to treatment at Week 12 in Part 1 receive second regimen of intravesical administration of SCH 721015 with Syn3 on same Day 1 and Day 4 regimen at same dose level.
  Interventions: Drug: SCH 721015

INTERVENTIONS:
Drug: SCH 721015 — Intravesical SCH 721015 (on Day 1 and 4) at a dose concentration of 3x1011particles/mL given in a 75 mL total volume. Administered into bladder through a urinary catheter, 75 mL will be instilled, left in the bladder for 1 hour, plus or minus 10 minutes. During the dwell time, subject will be repositioned from left to right, back and abdomen to maximize bladder surface exposure, approximately every 15 minutes.
  Other Names: rAd-IFN

SUMMARY:
The goal of this part (Part 1) of this clinical research study is to learn about the safety of giving 2 doses of SCH 72105 (also known as rAd-IFN) directly into the bladder to patients with bladder cancer that has come back. The goal of Part 2 of this study is to learn about the safety of giving 2 more doses of SCH 72105 directly into the bladder of Part 1 participants who had no sign of bladder cancer after Week 12. The level of effectiveness of SCH 72105 will also be studied by measuring the interferon (IFN) levels in the urine.

DETAILED DESCRIPTION:
The Study Drug:

SCH 72105 is designed to cause "gene transfer" by giving a gene called interferon -alpha-2b into the body. SCH 72105 is made after being processed in the lab with a study drug called Syn3. This combination of study drugs is also called SCH 721015 with Syn3. Syn3 is designed to help the body make a protein called interferon -alpha-2b, and this may help the body's immune system to react against the cancer.

Study Drug Administration:

On Days 1 and 4, SCH 72105 will be given into your bladder over about 1 minute through a urinary catheter. A urinary catheter is a thin flexible tube placed through the urinary tube and into the bladder. SCH 72105 will stay in the bladder for about 1 hour. You will be asked to turn from left to right, back to stomach, every 15 minutes to allow the bladder surface to be exposed to the drug.

A belladonna and opium (B&O) suppository will be inserted into your rectum about 30 minutes before the study drug doses. Levsin SL (hyoscyamine sulfate) will be given by mouth about 15 minutes before the study drug doses. These drugs are used to lower the risk of urinary urgency (a strong need to urinate).

Study Visits:

On Day 1:

* Blood (about 3 teaspoons) will be drawn for routine tests.
* Urine will be collected to test for IFN levels and to check for infection.
* Your vital signs will be measured before and after the study drug dose.
* You will be asked about any side effects and urinary symptoms you may have had and any drugs you may be taking.
* Your performance status will be recorded.

On Days 2 and 3 and on Days 5-14:

* Urine will be collected for biomarker testing. Biomarkers in your urine may be related to your reaction to the study drug.
* Your performance status will be recorded.
* You will be asked about any side effects and urinary symptoms you may have had and any drugs you may be taking.

On Day 4:

* Blood (about 3 teaspoons) will be drawn for routine tests.
* Urine will be collected for biomarker testing and to check for infection.
* Your vital signs will be measured before and after the study drug dose.
* You will be asked about any side effects and urinary symptoms you may have had and any drugs you may be taking.
* Your performance status will be recorded.

During Days 1-11, you will add about 1/2 cup of bleach to the toilet bowl before every time you urinate. You will then wait 15 minutes before flushing. You should avoid public bathrooms on these days. This procedure is required to avoid exposing other people to the study drug.

One (1) time a week during Weeks 2-11, the study staff will call and ask you about any side effects and urinary symptoms you may have had and any drugs you may be taking. During these calls, your performance status will also be recorded.

At Week 12:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* Urine will be collected for biomarker testing and to check for infection.
* Your vital signs will be measured.
* You will have an ECG. This ECG will be used as a screening test to help the doctor decide if you are eligible to take part in Part 2 of the study.
* Your performance status will be recorded.
* You will be asked about any side effects and urinary symptoms you may have had and any drugs you may be taking.
* You will have a cystoscopy with biopsies to check the status of the disease. All areas that the doctor thinks might have a tumor will be biopsied. Your bladder will also be measured during this procedure.

Length of Participation:

You may receive the 2 doses of the study drug as planned, if the doctor thinks it is in your best interest. You will not be able to receive the second dose of the study drug if the disease gets worse or intolerable side effects occur.

Part 2 of the Study:

If the disease has completely responded by Week 12 (no sign of cancer), you will be asked to take part in Part 2 of this study. In Part 2, participants will receive another 2 doses of the study drug. There is a separate informed consent form that describes Part 2, including screening tests that will help the doctor decide if you are eligible. You will be asked to sign the informed consent form if you agree to take part.

The level of effectiveness of SCH72105 treatment will be studied by measurement of IFN levels in the daily urine collections.

End-of-Study Visit:

You may choose to stop your study participation at any time. If you choose to stop before the Week 12 visit, you will be asked to return for an end-of-study visit. You will also be called by the study staff to ask about your health 1 time a year for the next 2 years. The following tests and procedures will be performed at the end-of-study visit:

* You will have a physical exam.
* You will have an ECG.
* Urine will be collected for routine tests.

Follow-Up:

If you had any signs of bladder cancer at Week 12, the study staff will call you at Months 6, 9, 12, 24, and 36. You will be asked if you have had any serious side effects.

This is an investigational study. SCH 72105 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 9 patients will take part in this study (9 total, for Parts 1 and 2). All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing to give written informed consent and be able to adhere to dose and visit schedules.
2. Histologically proven recurrent urothelial carcinoma of the bladder or prostatic urethra, Stage Tis, Ta
3. Patients with recurrent T1 disease who do not wish to have cystectomy.
4. Subjects must have failed at least two prior courses of BCG with or without recombinant interferon alpha administration or be BCG intolerant. This includes either two six week induction courses of BCG or a 6 week induction course followed by a 3 week mini-induction course of maintenance BCG.
5. At least 3 months must have passed since last BCG therapy or intravesical treatment for bladder carcinoma.
6. Subjects must be 18 years of age or older
7. Life expectancy of at least 3 months
8. Adequate performance status (Karnofsky score >/= 70%)
9. Adequate laboratory values. a) Hemoglobin >/=10 gm/dL. b) White blood cell count (WBC) >/= 3000/µL. c) Absolute neutrophil count (ANC) >/= 1500/µL. d) Platelet count >/=100,000/µL. e) PT </= 1.5 x upper limit of normal (ULN). f) Activated partial thromboplastin time (aPTT) </= 1.5 x ULN. g) AST </=1.5 x ULN. h) ALT </= 1.5 x ULN. i) Total bilirubin </= 1.5 x ULN. j) Creatinine </=1.5 x ULN.
10. Female subjects of childbearing potential (Female subjects who are not surgically sterilized, not at least 1 year postmenopausal) must agree to use adequate contraception (e.g. intrauterine device (IUD), condom plus spermicide, diaphragm, or cervical cap plus spermicide) or medical contraception: during the study and for at least 1 month prior to drug administration and for 4 months after treatment. Females who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the Study.
11. Male subjects who are sexually active must agree to use a condom from the beginning of treatment and for 1 month after the last dose

Exclusion Criteria:

1. Pregnant or nursing women
2. Suspected hypersensitivity to interferon alpha
3. Participation in another clinical trial or use of any investigational drug within 30 days prior to study entry
4. Subjects with organ transplants
5. Any known preexisting medical condition that could interfere with the subject's participation in and completion of the study such as:
6. b. Central nervous system (CNS) trauma or active seizure disorders requiring medication
7. c. Significant cardiovascular dysfunction within the past 6 months including symptomatic cardiac ischemia, arrhythmia or congestive heart failure requiring hospitalization or emergency room visit within last 3 months
8. d. Poorly controlled diabetes mellitus (HbA1C >10.0%);
9. e. Unstable pulmonary disease requiring hospitalization or emergency room visit within the last 3 months.
10. f. Immunologically mediated disease (eg, rheumatoid arthritis, autoimmune hepatitis, immune mediated glomerulonephritis).
11. Donation of blood within the preceding 60 days prior to study registration.
12. Any other condition that, in the opinion of the investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the protocol.
13. History of any clinically significant local or systemic infectious disease within 4 weeks prior to initial treatment administration
14. Untreated bladder infection
15. Positive for hepatitis BsAg or HIV Ab or hepatitis C
16. Immunosuppressive therapy within the last 3 months
17. Subjects who are part of the staff personnel directly involved with this study
18. Subjects who are family members of the investigational study staff
19. Traumatic catheterization within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety + Tolerability of 2 Instillations of Intravesical SCH 721015 in Admixture with Novel Excipient SCH 209702 (Syn3) on Day 1 and Day 4 | Daily urine collection for 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Colin P. Dinney, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org